CLINICAL TRIAL: NCT02218294
Title: A Phase 1 Study to Evaluate the Absorption, Metabolism and Excretion of BCX4161 Following Administration of a Single, Oral Dose of [14C]-Radiolabelled BCX4161 to Healthy Male Subjects
Brief Title: Study to Determine How BCX4161 is Metabolized and Eliminated by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX4161-103
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Hereditary Angioedema
Keywords: BCX4161; BioCryst; hereditary angioedema; mass balance; kallikrein inhibitor; ADME
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — avoralstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C] BCX4161 (Experimental): Includes a radiolabelled dose of [14C] BCX4161 and unlabelled BCX4161
  Interventions: Drug: BCX4161

INTERVENTIONS:
Drug: BCX4161

SUMMARY:
The purpose of the study is to assess the extent that radioactive dose of BCX4161 taken by mouth ends up in the urine, feces and expired air. If there are metabolites of BCX4161 made by the body, the chemical composition of these metabolites and their profile over time in blood and urine will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age 30 to 65 years of age (inclusive)
3. Body mass index of 18.0 to 32.0 kg/m2
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. A history of regular bowel movements
7. Must agree to use an adequate method of contraception

Key Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months
2. Current or history of any drug or alcohol abuse in the past 2 years or positive drugs of abuse screen
3. Current smokers
4. Radiation exposure, including that from the present study, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years
5. Clinically significant medical history, current medical or psychiatric condition, ECG finding, or laboratory/urinalysis abnormality
6. Activated partial thromboplastin time or PT outside of normal laboratory limits

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mass balance of BCX4161 after a single oral dose of [14C] BCX4161 based upon radioactivity excreted in urine, expired air and feces | Determined from samples drawn up to 14 days post-dose

SECONDARY OUTCOMES:
Chemical structure elucidation of major metabolites of [14C] BCX4161 in urine, plasma, feces, urine | Determined from samples drawn up to 4 days post-dose
Plasma pharmacokinetics (Cmax, Tmax, Tlag, AUC(0-last), AUC(0-inf), CL/F, Vz/F, AUC%extrapolated,t1/2, as applicable for each analyte) of total radioactivity, BCX4161, [14C] BCX4161 and major metabolites of [14C] BCX4161 | Data generated from samples drawn up to 7 days post-dose
Urinary pharmacokinetics (CLr, Ae, and % dose excreted) of BCX4161 | Data generated from samples drawn up to 7 days post-dose
Safety and tolerability evaluated through assessments of adverse events, laboratory analyses, vital signs, ECGs, and physical examinations | Over the duration of the study, approximately 6 weeks from screening through follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Collier, MBChB, FFPM, Dip Stats (OU), Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical Ltd, Ruddington, Nottingham, United Kingdom